CLINICAL TRIAL: NCT00662350
Title: Temperature Mapping of the Prostate With the Wallterm™ System
Acronym: WT-DK-TMW08
Status: Completed | Type: Observational
Sponsor: Pnn Medical A/S (Industry)
Responsible Party: Jacob Hyllested-Winge, M.D., VP, Director Clinical And Regulatory, Pnn Medical
Other Study IDs: WT-DK-TMW08
Record Dates: First submitted 2008-04-07; First posted 2008-04-21 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2010-02

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: BPH
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Symptomatic Benign Protate Hypertrophy: Symptom Score (IPSS) greater than 15, requiring invasive treatment, Prostate size greater than 25 g, Prostatic urethra length between 2.0 cm and 5.5 cm
  Interventions: Device: The Wallterm™ System

INTERVENTIONS:
Device: The Wallterm™ System — The Wallterm™ System is intended to ablate prostatic glandular and stromal tissue to relieve moderate to severe symptoms of outflow obstruction secondary to benign prostatic hyperplasia (BPH).
  Other Names: Wallterm™ Catheter (model 3010); Wallterm™ Central Unit (model 3020-10)

SUMMARY:
To measure intra-prostatic temperatures and evaluate the shape and size of necrotic lesions achieved under the standard treatment protocol in men with benign prostatic hyperplasia (BPH).

DETAILED DESCRIPTION:
The Wallterm System provides minimally invasive treatment of benign prostatic hyperplasia (BPH) via a high temperature, liquid filled, balloon thermotherapy. The catheter is composed of a silicone positioning balloon which anchors the catheter against the bladder neck. The multi-layer silicone treatment balloon may be adjusted to fit short (20-35mm) and long (40-55mm) prostates and is inflated (to approximately 650-700 mmHg / 20-22mm diameter) to ensure tight tissue contact and reduced blood perfusion. The handle contains the heating element and the liquid circulation mechanisms

ELIGIBILITY:
Inclusion Criteria:

* Men with symptomatic BPH requiring treatment,
* IPSS score > 15
* Age > 50 years
* Prostate size of 25 g or greater
* Prostatic urethra length between 2.0 cm and 5.5 cm,
* Ability to understand and consent to participate in this investigation,
* Willingness and ability to participate in all required follow-up evaluations.

Exclusion Criteria:

* Allergy towards Silicone,
* Peak Urinary Flow > 15 mL/s,
* Penile or urinary sphincter implant,
* Patients with active urinary tract infection indicated by a positive urinary culture >105 CFU (Note: These patients may be treated after successful treatment of the infection.)
* Clinical (historical), paraclinical (i.e. PSA> 10ng/mL) or histological evidence of prostatic cancer or bladder cancer,
* Evidence of a non-symmetric prostatic median lobe enlargement, or a prostatic lobe which is prominent with an obstructing "ball valve", as determined by cystoscopy or ultrasound,
* Patients with any previous prostate surgery, procedure for BPH, or any other invasive treatment to the prostate (such as TUR-P).
* Previous rectal surgery (Exception: hemorrhoid surgery), radical pelvic surgery or pelvic irradiation.
* Patients with confirmed or suspected bladder cancer.
* Patients with a history of cystolithiasis or bladder pathology, or who have experienced relapsing bacterial prostatitis within the last 6 months.
* Patients with gross haematuria. (Note: These patients may be eligible for this investigation if the results of a careful workup for cancer, including an X-ray study, cystoscopy and cytology, are found to be negative.)
* Patients with a history of bladder neck contracture.
* Patients who presently have urethral strictures, which prevent the passage of a 20 Fr endoscope (these patients may be treated after successful treatment of the stricture).
* Patients with neurogenic bladder dysfunction (neurogenic detrusor hypo- or hyperactivity).
* Patients interested in future fertility.
* Patients who have chronic catheter drainage due to urinary retention (these patients may be treated if a CMG demonstrates that the patient has a contractile bladder).
* Patients with bleeding disorders, or other systemic disorder contraindication minimally invasive surgical therapies.
* Any condition (ie: vascular clips) which would preclude an MRI from being performed, or otherwise confound this investigation.
* Patients with compromised renal function (i.e. serum creatinine >150 mls/l), renal or upper tract dilatation.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with BPH
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2008-06; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
To assess the temperatures within the prostate using the Wallterm System | Assessed at primary treatment

SECONDARY OUTCOMES:
To assess whether the Wallterm System delivers safe and consistent temperatures from base to apex; and determine the temperature range toward rectum, along the urethra. | Immediate
Delineate the extent and the location of necrosis | Short term

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen Nordling, Professor, Principal Investigator — Urological Dep., Herlev Hospital, Denmark
Locations (1):
- Herlev Hospital, Herlev, Denmark